CLINICAL TRIAL: NCT02019056
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled,Phase 2 Study to Evaluate the Efficacy, Safety of MG in Patients With Alcoholic Fatty Liver Disease and Alcoholic Hepatitis
Brief Title: Efficacy and Safety of MG in the Patients With Alcoholic Fatty Liver Disease and Alcoholic Hepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaKing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MG
Record Dates: First submitted 2013-10-30; First posted 2013-12-24 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Alcoholic Fatty Liver Disease; Alcoholic Hepatitis
MeSH Terms: conditions — Fatty Liver, Alcoholic; Hepatitis, Alcoholic | interventions — metadoxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): enteric coated capsule
  Interventions: Drug: Placebo /bid P.O
- MG 500mg (Experimental): Metadoxine + garlic oil
  Interventions: Drug: MG-1
- MG 1000mg (Experimental): Metadoxine + garlic oil
  Interventions: Drug: MG-2 : MG1000mg, Placebo /bid P.O
- Metadoxine 500mg (Sham Comparator): enteric coated capsule
  Interventions: Drug: metadoxine

INTERVENTIONS:
Drug: Placebo /bid P.O
  Arms: Placebo
Drug: MG-1
  Other Names: MG500mg,Placebo /bid P.O
  Arms: MG 500mg
Drug: MG-2 : MG1000mg, Placebo /bid P.O
  Arms: MG 1000mg
Drug: metadoxine
  Other Names: placebo, metadoxine 500mg/ bid P.O
  Arms: Metadoxine 500mg

SUMMARY:
The Purpose of A Multicenter, Randomized, Double-blind, Placebo-controlled to Evaluate the Efficacy, Safety and Pharmacokinetics of MG in Patients With alcoholic Fatty Liver Disease and Alcoholic Hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* •Patients over 18, under 70 years of age

  * The chronic alcohol intake patients

    * Current the heavy drinker over 3month, Day the average alcohol consumption Male>=60g, Female>=40mg y-GTP increase Male>=75, Female>=35
  * Over 1.5 ratio of AST to ALT
  * Patients who have chronoc alcohol disease

Exclusion Criteria:

* Patients who have liver disease with the cause different with the alcohol except
* Patients who have pyridoxine allergy or history
* Patients who are judged by investigator that participation of the study is difficult due to disease as follow; hepatic cirrhosis, Wilson's disease, malignant tumor, serious metabolic disease, severe renal disease, severe pulmonary disease, severe cardiovascular disease, severe nervous disease/psychiatric disorder, muscle disease and etc
* Patients taking other investigational product within 90 days prior to the participation in the study.
* Patients who has been taken any medications that could affect the treatment : hypoglycemic agents, colchicine, penicillamine, corticosteroids, ursodeoxycholic acid, pentoxifylline, lont-term use of NSAIDs, statins, neuroleptics, anti convulsive medications, high-dose acetaminophen(>=2.5g/day)
* Patients who have received treatment that may affect liver function within 1 month prior to the participation in the study
* Patient who considered ineligible for participation in the study as Investigator's judgment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in AST at 14weeks | 14Weeks
  To evaluate the liver function to assess improvement of the MG on change in AST lab value assessed from baseline to 12 weeks in patients with Alcoholic fatty liver disease
Number of Participants with Adverse Events (Safety) | 14weeks
  Adverse Event: Physical examine, Lab test, Vital sign, ECG, symptom, start day and time, end day and time, severity, progress, outcome, relation with investigational product.
To evaluate ALT normalization | 14weeks
  To evaluate ALT normalization assessed by comparing the percentage.
To evaluate AST normalization | 14weeks
  To evaluate AST normalization assessed by comparing the percentage.
change in AST, ALT, total lab billirubin lab value | 14weeks
  To evaluate the efficacy of the MG on change in AST, ALT, total lab billirubin lab value assessed from baseline to 4, 8, 12 weeks in patients with Alcoholic fatty liver disease

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang university Hospital, Guri-si, Gyeonggi-do, South Korea